CLINICAL TRIAL: NCT01786265
Title: A Randomized Study of Finite Androgen Ablation vs. Finite Androgen Ablation in Combination With Abiraterone Acetate and Prednisone in Patients With Prostate Cancer Who Have PSA Progression After Prostatectomy and/or Radiotherapy
Brief Title: Finite Androgen Ablation With or Without Abiraterone Acetate and Prednisone in Treating Patients With Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0993; NCI-2018-01856 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0993 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; bicalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Flutamide; Salicylic Acid; Goserelin; Leuprolide; luprolide acetate gel depot; nilutamide; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (finite androgen ablation) (Active Comparator): Participants receive either leuprolide acetate via injection every month or every 4 months, goserelin acetate via injection every month, or degarelix via injection every month for 8 months. Patients also receive bicalutamide PO QD, flutamide PO TID, or nilutamide PO QD. Patients may crossover to Arm B with disease progression after 8 months.
  Interventions: Drug: Bicalutamide; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Drug: Nilutamide
- Arm B (finite androgen ablation, abiraterone, prednisone) (Experimental): Participants receive leuprolide acetate, goserelin acetate, degarelix, bicalutamide, flutamide, or nilutamide as in Arm A. Patients also receive abiraterone acetate PO daily for 8 months and prednisone daily. Patients may crossover to Arm A with disease progression after 8 months.
  Interventions: Drug: Abiraterone Acetate; Drug: Bicalutamide; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Drug: Nilutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
  Arms: Arm B (finite androgen ablation, abiraterone, prednisone)
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Degarelix — Given via injection
  Other Names: FE200486; Firmagon
Drug: Flutamide — Given PO
  Other Names: 4''-Nitro-3''-trifluoromethylisobutyranilide; Apimid; Cebatrol; Chimax; Cytomid; Drogenil; Euflex; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolide; Oncosal; Profamid; Propanamide, 2-Methyl-N-(4-nitro-3-(trifluoromethyl)phenyl)-; Prostacur; Prostadirex; Prostica; Prostogenat; Sch 13521; Tafenil; Tecnoflut; Testotard
Drug: Goserelin Acetate — Given via injection
  Other Names: ZDX; Zoladex
Drug: Leuprolide Acetate — Given via injection
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Nilutamide — Given PO
  Other Names: Anandron; Nilandron; RU-23908
Drug: Prednisone
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm B (finite androgen ablation, abiraterone, prednisone)

SUMMARY:
This phase II trial studies how well finite androgen ablation with or without abiraterone acetate and prednisone work in treating patients with prostate cancer that has come back. Androgen can cause the growth of prostate cancer cells. Hormone therapy, such as finite androgen ablation, using leuprolide acetate, goserelin acetate, degarelix, bicalutamide, flutamide, and nilutamide may fight prostate cancer by lowering the amount of androgen the body makes. Abiraterone acetate may help to decrease the production of testosterone, and prednisone may help lower or prevent some side effects. It is not yet known whether giving acetate, goserelin acetate, degarelix, bicalutamide, flutamide, and nilutamide with or without abiraterone acetate and prednisone may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether finite maximal androgen ablation (8 month), as compared to luteinizing-hormone-releasing hormone (LHRH) alone, will improve one-year post-treatment prostate specific antigen (PSA)-free survival by 20%.

SECONDARY OBJECTIVES:

I. To determine testosterone recovery difference between the two groups. II. Calculate the PSA-free survival following testosterone recovery. III. To determine in the steroid biosynthesis metabolome, in the blood and bone marrow of patients at baseline, maximum response (eight months therapy) and upon PSA progression, evidence of minimal residual cancer (MD Anderson Cancer Center [MDACC] main campus patients only).

IV. To apply technologies in development able to detect presence of cancer cells ("minimal residual disease") at a clinical study milestone (baseline, completion of therapy and upon PSA progression).

EXPLORATORY OBJECTIVE:

I. To explore in archival tissue samples for a candidate predictive signature of outcome applying technologies for interrogation of protein deoxyribonucleic acid (dna) and ribonucleic acid (rna) levels of molecular markers / pathways of interest.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive either leuprolide acetate via injection every month or every 4 months, goserelin acetate via injection every month, or degarelix via injection every month for 8 months. Patients also receive bicalutamide orally (PO) once daily (QD), flutamide PO three times daily (TID), or nilutamide PO QD. Patients may crossover to Arm B with disease progression after 8 months.

ARM B: Patients receive leuprolide acetate, goserelin acetate, degarelix, bicalutamide, flutamide, or nilutamide as in Arm A. Patients also receive abiraterone acetate PO daily for 8 months and prednisone daily. Patients may crossover to Arm A with disease progression after 8 months.

After completion of study treatment, patients are followed up every 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document indicating that the subjects understand the purpose of and procedures required for the study and are willing to participate in the study
* Written Authorization for Use and Release of Health and Research Study Information has been obtained
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Life expectancy >= 12 months
* ECOG performance status (PS) =< 2
* Histologically documented diagnosis of adenocarcinoma of the prostate (PCa) with no histologic variants
* Prostate cancer recurrence after definitive local therapy (radical prostatectomy and/or radiation therapy) as evidenced by rising serum PSA, without evidence of metastases by bone scan or computed tomography (CT) scan

  * After radiation: A rising PSA taken to indicate recurrent prostate cancer in patients with previous definitive external beam radiotherapy will be defined as PSA of 1.0
  * After Radical Prostatectomy: A rising PSA taken to indicate recurrent prostate cancer in patients with previous radical prostatectomy will be defined by the criteria of the American Urological Association as any PSA measurement of 0.2, with a subsequent measurement > 0.2 ng/mL
* Patients who have received androgen ablative therapy for less than 8 weeks immediately prior to initiation of study drug are eligible provided they had only PSA evidence of progression (as defined above) with no visible metastases by CT-scan and bone scan (within 6 weeks) prior to starting androgen ablation
* White blood cell (WBC) >= 3.5 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x the upper limit of normal
* Serum potassium of >= 3.5 mEq/L
* Serum albumin of >= 3.0 g/dL
* Serum creatinine =< 1.5 x ULN
* Patients must have recovered from prior treatment regimens, e.g. surgery, radiation
* A patient who is sexually active and their partner must agree and use two reliable barrier forms of contraception (for example, condoms and diaphragm), from first day of study drug administration until for 1 week after last dose of abiraterone acetate, unless partner is post-menopausal
* Able to swallow the study drug whole as a tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken

Exclusion Criteria:

* Patients who have received prior hormonal therapy are excluded from the trial, except for: patients who have received up to 6 months of hormonal therapy as neoadjuvant therapy before radical prostatectomy or while on radiation therapy, as long as more than 1 year has elapsed between discontinuation of the neoadjuvant hormonal therapy and initiation of hormonal treatment for relapsing disease
* Any known metastases
* Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (>= 450 msec)
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
* Significant co-morbidity that could affect the safety or evaluability of participants as assessed by the treating physician and or principal investigator
* Prior therapy with strontium-89, samarium, rhenium-186 etidronate, chemotherapy or androgen biosynthesis inhibitors for prostate cancer is not allowed. Previous immunologic, homeopathic, natural, or alternative medicine therapies are acceptable provided treatment ended greater than 28 days prior to initiation of study drug
* Patients who, in the opinion of the investigator, are unable to comply with the requirements of the study protocol are not eligible
* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Active or symptomatic viral hepatitis
* History of pituitary or adrenal dysfunction
* Administration of an investigational therapeutic drug within 30 days of cycle 1 day 1
* Have known allergies, hypersensitivity, or intolerance to abiraterone acetate or prednisone or their excipients
* Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Have a pre-existing condition that warrants long-term corticosteroid use in excess of study dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2013-02-05 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) free survival (PSA < 0.1 ng/ml) | At 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org